CLINICAL TRIAL: NCT01780779
Title: Osteosarcoma and Ewing Sarcoma Treatment Response Assessment With Functional MRI Imaging in Children and Young Adults
Acronym: FUBEO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Steven Pans, Medical Doctor Radiologist, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: FUBEO; S51516 (Other: Ethical Committee Univ.Hospital)
Record Dates: First submitted 2013-01-23; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Ewing Sarcoma; Osteosarcoma
Keywords: Diffusion weighted MRI; Patient outcome assessment; Treatment response; Histopathology
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Osteosarcoma: All patients with Osteosarcoma), proven by surgical biopsy and histopathology.
  All included patients will be treated by chemotherapy (EURAMOS protocol)
  An MRI will be performed before, during and post-treatment
  Interventions: Other: MRI
- Ewing Sarcoma: All patients with proven diagnosis of Ewing sarcoma, proven by surgical biopsy and histopathology.
  All included patients will be treated by chemotherapy (EURO-EWING protocol)
  An MRI will be performed in all included patients before, during and after the chemotherapy
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI exam will be performed in all patients included in the study. The patients will be treated by chemotherapy, defined in the EURO-EWING or EURAMOS protocol.
  The MR findings will not have any impact on the treatment.

SUMMARY:
The purpose of the study was to investigate whether functional MRI imaging (diffusion weighted imaging) is useful for monitoring the therapeutic response of bone sarcomas in children and young adults. All patients will be scanned before, during and after chemotherapy. The findings on MRI will be correlated with histological finding after surgery.

Second purpose : to define apparent diffusion coefficient value of the bone sarcoma.

Third purpose : to try define prognostic factors, to investigate if there is a correlation between early treatment response and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ewing or Osteosarcoma, proven by biopsy and histopathology
* all patients are treated by chemotherapy defined by EURAMOS and EURO-EWING protocol

Exclusion Criteria:

* Patients under the age of 6 years old
* patients with contra-indication for MR exam (pace-maker...)
* Patients with renal insufficiency
* Claustrophobia

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with Ewing sarcoma or Osteosarcoma, proven by biopsy and histolopathology.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
tumor necrosis - therapy response | 6 months
  correlation of MRI findings with clinical findings during chemotherapy correlation of diffusion weighted MRI and histopathology results after surgical resection.
  Calculation of apparent diffusion coefficient : is it a valuable parameter?

SECONDARY OUTCOMES:
Prognosis and outcome | 2 years
  Is there a correlation between early treatment response and outcome? Is diffusion weighted MRI able to predict outcome of the patient (prognostic factor)?

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium